CLINICAL TRIAL: NCT05953194
Title: Effects of Anti-sugar-sweetened-beverage Counter-marketing on Behavioral Intentions and Perceived Weight Stigma
Brief Title: Effects of Sugary Drinks Counter-marketing Messages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Harvard Pilgrim Health Care (Other)
Responsible Party: Principal Investigator, Anna Grummon, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 69580a
Record Dates: First submitted 2023-07-11; First posted 2023-07-20 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Obesity; Weight Prejudice; Weight Gain; Dietary Habits
Keywords: counter-marketing; health communication; sugar sweetened beverage
MeSH Terms: conditions — Obesity; Weight Prejudice; Weight Gain; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (neutral) messages (Active Comparator): Participants will view control messages approximately matched to the intervention messages on length, but discussing a neutral topic unrelated to sugary drinks (safe driving). Participants will view a total of 4 messages developed for this arm.
  Interventions: Behavioral: Exposure to control (neutral) messages
- Traditional health messages (Experimental): Participants will view traditional health messages focused on the health consequences of sugar-sweetened beverage consumption, using text adapted from prior sugary drink campaigns. Participants will view a total of 4 messages developed for this arm.
  Interventions: Behavioral: Exposure to traditional health messages
- Counter-marketing messages (Experimental): Participants will view counter-marketing messages about sugary drinks that incorporate principles of effective counter-marketing campaigns, including describing industry manipulation of consumers, appealing to emotions (especially anger), describing health consequences, and criticizing the industry for demographic targeting. Messages include text adapted from prior counter-marketing campaigns. Participants will view a total of 4 messages developed for this arm.
  Interventions: Behavioral: Exposure to counter-marketing messages

INTERVENTIONS:
Behavioral: Exposure to counter-marketing messages — Counter-marketing messages about sugary drinks that incorporate principles of effective counter-marketing campaigns, including describing industry manipulation of consumers, appealing to emotions (especially anger), describing health consequences, and criticizing the industry for demographic targeting. Messages include text adapted from prior counter-marketing campaigns. Participants will view a total of 4 messages developed for this arm.
  Arms: Counter-marketing messages
Behavioral: Exposure to traditional health messages — Traditional health messages focused on the health consequences of sugar-sweetened beverage consumption, using text adapted from prior sugary drink campaigns. Participants will view a total of 4 messages developed for this arm.
  Arms: Traditional health messages
Behavioral: Exposure to control (neutral) messages — Control messages approximately matched to the intervention messages on length, but discussing a neutral topic unrelated to sugary drinks (safe driving). Participants will view a total of 4 messages developed for this arm.
  Arms: Control (neutral) messages

SUMMARY:
This study aims to examine consumer responses to traditional and counter-marketing messages discouraging sugary drink consumption, including effects on intentions to consume sugary drinks and perceived weight stigma. Because prior research has suggested that counter-marketing may be especially effective among younger populations, the investigators will examine effects overall and by age group (young adults [ages 18-29 years] vs. middle and older adults [ages 30+ years]).

DETAILED DESCRIPTION:
In this online randomized clinical trial, participants will be randomized to one of three arms: 1) Control (neutral) messages, 2) Traditional health messages, and 3) Counter-marketing messages. In each arm, participants will view four messages developed for their randomly assigned arm and answer questions about the messages and their behavioral intentions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older

Exclusion Criteria:

* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2184 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Intentions to consume sugary drinks | The survey will take up to 20 minutes
  We will assess intentions to consume sugary drinks using 2 items: "In the next week, I plan to drink sugary drinks like sodas, sports drinks, or fruit drinks," and "In the next week, I am likely to drink sugar-sweetened beverages like sodas, sports drinks, or fruit drinks". Response options to both items will use a 5-point Likert scale: the first item's response options will range from "definitely not" (1) to "definitely yes" (5), and the second item's response options will range from "not at all likely" (1) to "extremely likely" (5). We will average responses to the 2 items.

SECONDARY OUTCOMES:
Perceived message effectiveness for discouraging sugary drink consumption | The survey will take up to 20 minutes
  Item: "These messages discourage me from wanting to drink sugary drinks." This variable will be measured on a 5-point Likert scale ranging from "not at all" (1) to "a great deal" (5).
Negative feelings toward drinking sugary drinks | The survey will take up to 20 minutes
  Item: "How do these messages make you feel about drinking sugary drinks?" This variable will be measured on a 5-point Likert scale ranging from "extremely positive" (1) to "extremely negative" (5).
Anticipated social interactions | The survey will take up to 20 minutes
  We will examine anticipated social interactions by asking, "How likely are you to talk about these messages with others in the next week?" This item will be scored on a 5-pt Likert scale ranging from "not at all likely" (1) to "extremely likely" (5).
Attitudes toward sugary drink companies | The survey will take up to 20 minutes
  We will examine attitudes toward sugary drink companies by asking, "How do you feel about companies that make sugary drinks?" This item will be scored on a 5-pt Likert scale ranging from "dislike them a lot" (1) to "like them a lot" (5).
Perceived obesity stigma | The survey will take up to 20 minutes
  We will examine the extent to which participants perceive the messages as contributing to obesity stigma by asking 3 items: "These messages promote negative attitudes about people who have overweight or obesity," "These messages increase blame towards people for being overweight," and "These messages make obesity seem like a much simpler issue than it really is." Each item will be scored on a 5-point Likert scale from "not at all" (1) to "a great deal" (5). We will average responses to these items.
Message reactance | The survey will take up to 20 minutes
  We will examine psychological reactance to the messages by asking 3 items: "These messages are trying to manipulate me," "These messages are overblown" and "How much do these messages make you feel angry?" Each item will be scored on a 5-point Likert scale from "not at all" (1) to "a great deal" (5). We will average responses to these items, assuming sufficient internal consistency (alpha>=.70).

CONTACTS AND LOCATIONS:
Overall Officials: Anna H Grummon, PhD, Principal Investigator — Stanford School of Medicine, Department of Pediatrics
Locations (1):
- Stanford School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share statistical analysis plan and analytic code after publication. The investigators will post these items and de-identified data on ResearchBox, a publicly available platform.
Supporting Information: SAP, Analytic Code
Time Frame: Within 6 months of publication
Access Criteria: There will be no access criteria; information will be publicly available. We plan to make these resources available on ResearchBox.
URL: http://researchbox.org

REFERENCES:
- [Background] Kraak VI, Consavage Stanley K, Harrigan PB, Zhou M. How have media campaigns been used to promote and discourage healthy and unhealthy beverages in the United States? A systematic scoping review to inform future research to reduce sugary beverage health risks. Obes Rev. 2022 May;23(5):e13425. doi: 10.1111/obr.13425. Epub 2022 Feb 9. PMID 35142020
- [Background] Boles M, Adams A, Gredler A, Manhas S. Ability of a mass media campaign to influence knowledge, attitudes, and behaviors about sugary drinks and obesity. Prev Med. 2014 Oct;67 Suppl 1:S40-5. doi: 10.1016/j.ypmed.2014.07.023. Epub 2014 Jul 24. PMID 25066020
- [Background] Kite J, Grunseit A, Bohn-Goldbaum E, Bellew B, Carroll T, Bauman A. A Systematic Search and Review of Adult-Targeted Overweight and Obesity Prevention Mass Media Campaigns and Their Evaluation: 2000-2017. J Health Commun. 2018;23(2):207-232. doi: 10.1080/10810730.2018.1423651. Epub 2018 Jan 16. PMID 29336684
- [Background] Te V, Ford P, Schubert L. Exploring social media campaigns against sugar-sweetened beverage consumption: A systematic search. Schumacher U, ed. Cogent Medicine. 2019;6(1):1607432. doi:10.1080/2331205X.2019.1607432
- [Background] Bryan CJ, Yeager DS, Hinojosa CP. A values-alignment intervention protects adolescents from the effects of food marketing. Nat Hum Behav. 2019 Jun;3(6):596-603. doi: 10.1038/s41562-019-0586-6. Epub 2019 Apr 15. PMID 30988478
- [Background] Crandall CS, Reser AH. Attributions and Weight-Based Prejudice. In: Brownell K, Puhl R, Schwartz M, Rudd L, eds. Weight Bias: Nature, Consequences, and Remedies. Guilford Publications; 2005:83-96.
- [Background] Puhl RM, Schwartz MB, Brownell KD. Impact of perceived consensus on stereotypes about obese people: a new approach for reducing bias. Health Psychol. 2005 Sep;24(5):517-25. doi: 10.1037/0278-6133.24.5.517. PMID 16162046
- [Background] Dixon H, Scully M, Gascoyne C, Wakefield M. Can counter-advertising diminish persuasive effects of conventional and pseudo-healthy unhealthy food product advertising on parents?: an experimental study. BMC Public Health. 2020 Nov 25;20(1):1781. doi: 10.1186/s12889-020-09881-1. PMID 33238936
- [Background] Krieger J, Kwon T, Ruiz R, Walkinshaw LP, Yan J, Roberto CA. Countermarketing About Fruit Drinks, Alone or With Water Promotion: A 2019 Randomized Controlled Trial in Latinx Parents. Am J Public Health. 2021 Nov;111(11):1997-2007. doi: 10.2105/AJPH.2021.306488. Epub 2021 Oct 28. PMID 34709859
- [Derived] Grummon AH, Zeitlin AB, Lee CJY, Hall MG, Collis C, Cleveland LP, Petimar J. Countermarketing Versus Health Education Messages About Sugar-Sweetened Beverages: An Online Randomized Controlled Trial of US Adults. Am J Public Health. 2024 Dec;114(12):1354-1364. doi: 10.2105/AJPH.2024.307853. Epub 2024 Oct 3. PMID 39361914